CLINICAL TRIAL: NCT02823457
Title: Evaluating Values-based Motivational Interviewing to Increase Treatment Completion With Fixed Dose Combination MK-5172/MK-8742 Among Veterans With Active Substance Use Disorders and Treatment-naïve Genotype 1 Chronic Hepatitis C
Brief Title: VBMI to Increase Treatment Completion With MK-MK-5172/MK-8742 Among Veterans With Active Substance Use Disorders Genotype 1 Chronic Hepatitis C
Acronym: VBMI SUD/HCV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: G.V. (Sonny) Montgomery VA Medical Center (U.S. Federal Agency)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Mary Jane Burton, Staff Physician, G.V. (Sonny) Montgomery VA Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 53635
Record Dates: First submitted 2016-07-01; First posted 2016-07-06 (Estimated); Results first posted 2021-01-12 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Patient Adherence, Chronic Hepatitis C, Alcohol-related Disorders
MeSH Terms: conditions — Patient Compliance; Hepatitis C, Chronic; Alcohol-Related Disorders

STUDY DESIGN:
Masking Description: open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VBMI intervention group (Other): All patients will receive a 12 week VBMI intervention to promote treatment completion
  Interventions: Behavioral: VBMI

INTERVENTIONS:
Behavioral: VBMI — 12 week values based motivational interviewing intervention with a licensed psychologist
  Other Names: Values Based Motivational Interviewing

SUMMARY:
This study implement a values-based motivational interviewing (VBMI) intervention to promote treatment completion with fixed dose combination (FDC) MK-5172/MK-8742 x 12 weeks among 30 Veterans with substance use disorder (SUD) and treatment naïve genotype 1 chronic hepatitis C virus (HCV) infection.

DETAILED DESCRIPTION:
The investigators will conduct a prospective study of 30 Veterans with treatment-naive genotype 1 chronic hepatitis C infection admitted to the Substance Abuse Residential Rehabilitation Treatment Program (SARRTP) at the G.V. (Sonny) Montgomery VA Medical Center. Enrolled veterans will be treated MK-5172/MI-8742 while receiving a 12 week values based motivational intervention to promote completion of HCV treatment. MK-5172/MK-8742 will be prescribed in accordance with the package insert.

ELIGIBILITY:
Inclusion Criteria:

1. Identified as having treatment-naïve genotype 1 chronic HCV infection; Veterans who are genotype 1a must have baseline NS5a resistance testing
2. Current resident of the SARRTP program
3. Willing to initiate treatment with FDC MK-5172/MK-8742 during SARRTP and up to 30 days post-discharge.
4. Willing to attend coordinated HCV treatment clinic visits and substance abuse aftercare visits every 2 weeks upon SARRTP discharge

Exclusion Criteria:

1. Contraindications for therapy with FDC MK-5172/MK-8742
2. Unable to provide written informed consent
3. Hepatocellular carcinoma or other medical condition precluding HCV treatment
4. Acute HCV infection
5. Prior treatment for chronic HCV
6. History of decompensated cirrhosis
7. Platelet count < 75 K/cmm and/or albumin < 3 grams/dL
8. Females and male sex partners of females who are pregnant, nursing and/or unwilling to use contraception
9. Patients infected with genotype 1a who have not undergone baseline NS5a resistance testing

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Burton, MD, Principal Investigator — G.V. (Sonny) Montgomery VAMC
Locations (1):
- GV Sonny Montgomery VAMC, Jackson, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Burton MJ, Voluse AC, Patel AB. Supporting direct acting antiviral medication adherence and treatment completion in a sample of predominantly rural veterans with hepatitis C and substance use disorders. Addict Sci Clin Pract. 2024 Jun 25;19(1):51. doi: 10.1186/s13722-024-00480-8. PMID 38918869

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | VBMI Intervention Group
Started | 20
Completed | 15
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | VBMI Intervention Group
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.0 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 17
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Treatment Completion
Description: Number of participants who completed treatment
Time Frame: 12 weeks after initiation treatment
Measure: Count of Participants; unit: Participants
Arm/Group | VBMI Intervention Group
Number analyzed (Participants) | 20
Participants | 15

2. Secondary Outcome: Sustained Virologic Response
Description: Number of participants who achieved SVR
Time Frame: an average of 3 months after treatment completion
Measure: Count of Participants; unit: Participants
Arm/Group | VBMI Intervention Group
Number analyzed (Participants) | 20
Participants | 19

ADVERSE EVENTS:
Time Frame: Six months
Arm/Group | VBMI Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-10): https://cdn.clinicaltrials.gov/large-docs/57/NCT02823457/Prot_SAP_000.pdf